CLINICAL TRIAL: NCT02381899
Title: Observational Study in Comorbid Patients With Chronic Lymphocytic Leukemia Receiving First-line Bendamustine With Rituximab
Brief Title: Observational Study in CLL Patients Receiving BR
Status: Completed | Type: Observational
Sponsor: Czech CLL Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: BR-1
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; bendamustine; rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BR in CLL: Patients receive bendamustine hydrochloride 90mg/m2 IV on days 1 and 2 each cycle. Patients also receive rituximab 375 mg/m2 IV on day 1 at first cycle and 500 mg/m2 on day 1 all subsequent cycles.
  Interventions: Drug: Bendamustine and Rituximab

INTERVENTIONS:
Drug: Bendamustine and Rituximab — Patients receive bendamustine and rituximab. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Mabthera; Levact

SUMMARY:
The purpose of this observational study is to provide additional data to confirm the safety profile and efficacy of bendamustine and rituximab (BR) chemotherapy for chronic lymphocytic leukemia patients with significant comorbidities treated in routine clinical practice.

DETAILED DESCRIPTION:
BR (bendamustine, rituximab) combination is currently accepted as a first-line treatment of chronic lymphocytic leukemia (CLL) in patients for whom fludarabine combination chemotherapy is not appropriate.

The objective of this observational study is to provide additional data to confirm the safety profile and efficacy of BR for CLL patients treated in routine clinical practice.

Specific data of interest are: comorbid conditions, CLL characteristics, adverse events, reasons for discontinuation BR, overall response rates, complete response rate, progression-free survival, overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic lymphocytic leukemia
* Patients treated with first-line BR for active disease requiring treatment
* Cumulative Illness Rating Scale (CIRS) > 6
* Informed consent to data collection

Exclusion Criteria:

* Patients treated with BR within prospective clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lymphocytic leukemia.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Toxicity assessed by Common Toxicity Criteria for Adverse Effects (CTCAE) criteria | 8 months
  Toxicity assessed by Common Toxicity Criteria for Adverse Effects (CTCAE) criteria (myelotoxicity, infections, etc.)
Overall response rate | 8 months
  Response to treatment was assessed using National Cancer Institute-sponsored Working Group criteria, including bone marrow examination and radiographic confirmation of complete response.

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Calculated from the start of therapy until disease progression or death
Overall survival | 3 years
  Time interval from the start of therapy until death form any cause

CONTACTS AND LOCATIONS:
Overall Officials: Martin Spacek, MD, PhD, Study Chair — Czech CLL Study Group
Locations (5):
- Czechia (5):
  - Department of Hematology - Oncology, University Hospital, Brno
  - 4th Department of Medicine - Hematology, University Hospital, Hradec Králové
  - Department of Hematology, University Hospital, Pilsen
  - Department of Medicine - Hematology, University Hospital Kralovske Vinohrady, Prague
  - 1st Department of Medicine - Hematology, General University Hospital, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer K, Cramer P, Busch R, Bottcher S, Bahlo J, Schubert J, Pfluger KH, Schott S, Goede V, Isfort S, von Tresckow J, Fink AM, Buhler A, Winkler D, Kreuzer KA, Staib P, Ritgen M, Kneba M, Dohner H, Eichhorst BF, Hallek M, Stilgenbauer S, Wendtner CM. Bendamustine in combination with rituximab for previously untreated patients with chronic lymphocytic leukemia: a multicenter phase II trial of the German Chronic Lymphocytic Leukemia Study Group. J Clin Oncol. 2012 Sep 10;30(26):3209-16. doi: 10.1200/JCO.2011.39.2688. Epub 2012 Aug 6. PMID 22869884
- [Result] Obrtlikova P, Spacek M, Doubek M, Hadrabova M, Panovska A, Svackova K, Trneny M. Bendamustine with rituximab (BR) is safe treatment option with high response rate for chronic lymphocytic leukemia in elderly patients with comorbidities. LEUKEMIA & LYMPHOMA 56(1SI): 151-153, 2015 [abstract #180].
- [Result] Spacek M, Obrtlikova P, Hadrabova M, Cmunt E, Karban J, Molinsky J, Simkovic M, Mocikova H, Mohammadova L, Panovska A, Novak J, Smolej L, Doubek M, Trneny M. Observational study in comorbid patients with CLL receiving first-line rituximab-bendamustine. XVII International Workshop on CLL, New York, May 12-15, 2017 [abstract #148]
- [Derived] Spacek M, Obrtlikova P, Hrobkova S, Cmunt E, Karban J, Molinsky J, Simkovic M, Mocikova H, Mohammadova L, Panovska A, Novak J, Trneny M, Smolej L, Doubek M. Prospective observational study in comorbid patients with chronic lymphocytic leukemia receiving first-line bendamustine with rituximab. Leuk Res. 2019 Apr;79:17-21. doi: 10.1016/j.leukres.2019.02.002. Epub 2019 Feb 15. PMID 30797139
- See also: Czech CLL Study Group — http://www.cll.cz